CLINICAL TRIAL: NCT05900076
Title: Technical Feasibility of the Cell-free DNA Test for Non-invasive Cytogenetic Analysis of Early Miscarriages Versus the Gold Standard Microarray
Brief Title: Technical Feasibility of the cfDNA Test for Non-invasive Cytogenetic Analysis of Early Miscarriages Versus the Gold Standard Microarray
Acronym: NICAEA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0080
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Spontaneous Miscarriage
Keywords: Cell-free DNA; spontaneous miscarriage; chromosomal abnormalities; cytogenetic analysis
MeSH Terms: conditions — Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: This group corresponds to patients who have just suffered a miscarriage and are undergoing curettage for the evacuation of the product of conception.
  Interventions: Diagnostic Test: Curettage for the evacuation of the product of conception

INTERVENTIONS:
Diagnostic Test: Curettage for the evacuation of the product of conception — The product of conception taken during the intervention will be recovered at Day 1

SUMMARY:
Among the 15% of couples who experience a spontaneous early miscarriage (SEM) during their pregnancy, approximately 2 to 5% will suffer from recurrent SEM. It is only after the third SM that they will be offered a workup to look for a predisposition to SEM. This workup does not currently include a search for foetal chromosomal abnormalities that could be considered causal for this event. These anomalies are responsible for approximately 50% of SEM and their detection could lead to an explanation for half of the couples currently without a diagnosis after a standard workup. The diagnosis of chromosomal abnormalities can be made by karyotype analysis or by Cytogenetic Microarray Analysis (CMA) on the product of conception. Unfortunately, karyotyping has a high failure rate due to poor cell culture of samples that are often degraded or of low quantity. The CMA is not always feasible due to the absence of analyzable feto-placental material linked to the use of a drug strategy for its elimination.

The study of cell-free DNA of syncytiotrophoblastic origin (cfDNA) circulating in the maternal plasma could be a solution as it is for non-invasive prenatal screening of trisomy 21. cfDNA is detectable from 6 to 8 weeks of amenorrhea and released in the maternal blood as long as placental tissue is present in the uterus, can be easily obtained by maternal venous sampling. If maternal blood sampling is performed before complete removal of the product of conception, then detection of foetal chromosomal abnormalities would be possible. Thus, if failure rates of CMA and cfDNA techniques are comparable, cfDNA could be preferred as it applies for miscarriages for whom no fetoplacental material can be obtained.

This study therefore proposes to compare the failure rates of the two technologies (CMA and cfDNA) for the detection of chromosomal abnormalities in recurrent SEM.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has suffered a miscarriage and requires a curettage to collect the product of conception
* Patient consenting to constitutional cytogenetic analysis on cfDNA and product of conception
* Patient of legal age
* Patient affiliated to a Social Security system.

Exclusion Criteria:

* Venous sampling impossible
* Miscarriage before 8 weeks of pregnancy (unusable cfDNA)
* Patient does not understand French
* Patient under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15% of couples will experience spontaneous miscarriage during their reproductive life. Women that will go to the ObGyn Emergency Department of our Hospital where spontaneous miscarriage will be confirmed and curettage decided will be eligible for inclusion. No additional criterion applies.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Failure rate of cfDNA compared to CMA | The outcome measure (failure rates of both techniques) will be assessed through study completion ; estimated 6 months after last inclusion.
  Failure rate of cfDNA compared to CMA Since the difference in failure rates between the two techniques (MCA and cfDNA) corresponds to a comparison of 2 proportions in a matched situation.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Femme-Mère-Enfant; service gynécologie/obstétrique, Bron, Rhône
  - Hopital Femme-Mère-Enfant; service médecine de la reproduction, Bron, Rhône

IPD SHARING:
Plan to Share IPD: No